CLINICAL TRIAL: NCT00582036
Title: Glucose Control In Hematopoetic Stem Cell Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study terminated due to lack of enrollment
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma Center for the Advancement of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Glucose Control; OCAST HR06-13
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2011-04-22 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Hyperglycemia; Hematopoietic Stem Cell Transplantation
Keywords: Hyperglycemia; Hematopoietic stem cell transplantation; Bone marrow transplant; High blood sugar
MeSH Terms: conditions — Hyperglycemia | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Regular Sliding Scale Insulin administration for hyperglycemia
  Interventions: Drug: Regular Insulin
- Arm 2 (Experimental): MiniMed Paradigm monitoring device for hyperglycemia
  Interventions: Device: Deployment of the MiniMed Paradigm monitoring device

INTERVENTIONS:
Drug: Regular Insulin — Use of sliding scale insulin as per Appendix 1
  Arms: Arm 1
Device: Deployment of the MiniMed Paradigm monitoring device — Automated insulin delivery system
  Arms: Arm 2

SUMMARY:
To determine whether intensive glucose control results in improved mortality and reduced hospital stay length by performing a randomized trial of intensive glucose management (blood glucose goal 110 mg/dl) using continuous IV insulin and glucose vs. non-intensive glucose management (goal 200 mg/dl)

DETAILED DESCRIPTION:
TO determine whether there are fewer infections, days without a fever, days on antibiotics given for an infection and time to marrow engraftment are improved by intensive glucose management; and to determine whether there is evidence of a reduction in measures of inflammation in patients randomized to intensive glucose management and whether reduction of inflammation is associated with outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18
* Must meet standard criteria for HSCT
* If patient is known diabetic at admit the may be maintained on home sulfonylurea and insulin if randomized to the conventional arm

Exclusion Criteria:

* If on intensive arm patient must stop all oral hyperglycemic meds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Selby, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was not satisfactory to study completion; study terminated early.
Groups:
- Arm 1: Regular Sliding Scale Insulin per the following >400mg/dl = 12 units 351-400mg/dl = 10 units 301-350mg/dl = 8 units 251-300mg/dl = 6 units 200-250mg/dl = 4 units <200 No insulin
- Arm 2: Baseline IV Insulin infusion begins with:
  >220mg/dl - Start at 2 units/hr 110-220mg/dl - Start at 1 unit/hr <110 - Monitor fingerstick before meals and at bedtime
  Sliding Scale IV Insulin adjustments based on:
  >201mg/dl - Increase by 2 units/hr 141-200mg/dl - Increase by 1 unit/hr 111-140mg/dl - Increase by 0.5 units/hr 81 - 110mg/dl - If blood glucose decreases by 15mg/dl or more, reduce drip by 25% 61-80mg/dl - Reduce infusion by 25% <60 Stop infusion
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 5 | 6
Completed | 5 | 5 (One patient withdrew consent)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (1) | 58 (2) | 59 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Secondary Outcome: Reduction of Infection
Time Frame: About 100 days
Reporting Status: Not Posted

2. Secondary Outcome: Reduced Length of In-hospital Stay
Time Frame: About 100 days
Reporting Status: Not Posted

3. Primary Outcome: Intensive Control of Glucose Effects on Mortality in Allogenic Hematopoietic Stem Cell Transplant (HSCT)
Time Frame: 100 days
Population: Due to early termination, data not analyzed
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

LIMITATIONS AND CAVEATS:
This study was terminated early due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No